CLINICAL TRIAL: NCT02067416
Title: Prospective Study To Validate The Predictive Value Of Mammostrat Score, DDR Score And TLE3 Gene When A Taxane-Based Chemo Agents Or Anthracycline-Based Chemo Agent Is Used In The Neo-Adjuvant Setting
Brief Title: PREDATOR: Neoadjuvant Gene Prediction for Breast Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding agent withdrew funding
Sponsor: Jenny C. Chang, MD (Other)
Collaborators: GE Healthcare (Industry); The Methodist Hospital Research Institute (Other)
Responsible Party: Sponsor-Investigator, Jenny C. Chang, MD, Methodist Cancer Center Director (Rodriguez no longer at MCC), The Methodist Hospital Research Institute
Organization: The Methodist Hospital Research Institute (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00007624; 0712-0127 (Other: HMRI IRB)
Record Dates: First submitted 2014-02-17; First posted 2014-02-20 (Estimated); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Breast Cancer
Keywords: neoadjuvant; mammostrat; TLE3; DDR; breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Doxorubicin; Epirubicin; Paclitaxel; Docetaxel; Albumin-Bound Paclitaxel; ixabepilone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- taxane-based chemotherapy (Active Comparator): physician choice: taxane-based chemotherapy to include Paclitaxel, Docetaxel, Abraxane or Ixabepilone given as standard of care
  Interventions: Drug: taxane-based chemotherapy
- anthacycline based chemotherapy (Active Comparator): Physician choice: anthracycline based chemotherapy including Adriamycin, Epirubicin give as standard of care
  Interventions: Drug: Anthracycline based chemotherapy

INTERVENTIONS:
Drug: Anthracycline based chemotherapy — standard of care neoadjuvant treatment with anthracycline based chemotherapy
  Other Names: Adriamycin; Epirubicin
  Arms: anthacycline based chemotherapy
Drug: taxane-based chemotherapy — neoadjuvant taxane based chemotherapy given as standard of care
  Other Names: Paclitaxel; Docetaxel; Abraxane; Ixabepilone
  Arms: taxane-based chemotherapy

SUMMARY:
Study of the assay, Mammostrat®. to verify its utility as a predictor or outcome tool to determine whom would benefit from chemotherapy prior to surgery. Also could be used as a clinical marker to identify patients with breast cancer who do not benefit from some preoperative chemotherapies.

DETAILED DESCRIPTION:
The purpose of this phase II study is to find out if the test, Mammostrat® can be used as a predictor or outcome tool to determine who will best benefit from chemotherapy prior to surgery. This can be used to determine if Mammostrat assay may be used as a clinical marker to identify a subset of women with breast cancer who do not benefit from preoperative chemotherapy, either taxane/taxane-like (T) chemo agents or anthracycline-based chemotherapy and cyclophosphamide (AC).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologic confirmation of invasive breast carcinoma.
2. Patients must have intact primary tumor.
3. ≥18 years of age.
4. Patients with bilateral breast cancer are eligible.
5. Patients with second primary breast cancers are eligible.
6. The primary breast tumor must be ≥ 2 cm by physical exam or imaging.
7. The tumor must have been determined to be HER2-negative as follows:

   * Fluorescent in situ hybridization (FISH)-negative (defined by ratio of HER2 to CEP17 must be < 2.2)
   * Immunohistochemistry (IHC) 0-1+; or
   * IHC 2+ and FISH-negative
8. ECOG PS of 0, 1, or 2.
9. Negative serum pregnancy test ≤7 days of treatment initiation and a serum or urine pregnancy test must be repeated ≤ 3 days prior to starting treatment for women of childbearing potential (WOCBP). For WOCBP, adequate contraception must be used throughout the study. For this study, acceptable methods of contraception include a reliable intrauterine device or a spermicide in combination with a barrier method. Women who are already on hormonal forms of birth control may continue that treatment but must also use a barrier method.
10. Ability to understand the requirements of the study, provide written informed consent and authorization of use and disclosure of protected health information, and agree to abide by the study restrictions and return for the required assessments.
11. Patient must be willing to undergo breast biopsies as required by the study protocol.
12. Sufficient tissue must be available from the diagnostic core biopsies. If not, patients must undergo additional biopsies to perform Mammostrat.

Exclusion Criteria:

1. Patients with a history of other invasive malignancies diagnosed and treated within the previous 5 years, except non-melanoma skin cancer and non-invasive cervical cancer.
2. Prior treatment with any investigational drug within the preceding 4 weeks.
3. Evidence of New York Heart Association class III or greater cardiac disease.
4. History of myocardial infarction, stroke, ventricular arrhythmia, or symptomatic conduction abnormality within 6 months.
5. Concurrent severe or uncontrolled medical disease (i.e., active systemic infection, diabetes, hypertension, coronary artery disease, congestive heart Failure or major surgery) that, in the opinion of the Investigator, would compromise the safety of the patient or compromise the ability of the patient to complete the study.
6. Pregnant or nursing women.
7. Known allergic reaction to Cremophor or any of the chemo agents on this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-07; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Compare Mammostrat score clinical response rates to chemotherapy | 2 years
  The percentage of patients undergoing chemotherapy who have Mammostrat low risk scores will be calculated

SECONDARY OUTCOMES:
pathological complete response rate compare to predictors | 2 years
  The percentage of patients undergoing chemotherapy who have Mammostrat low risk scores will be calculated

CONTACTS AND LOCATIONS:
Overall Officials: Angel A Rodriguez, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Houston Methodist Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Cancer-related options for clinical trial participation — https://www.houstonmethodist.org/research/clinical-trials/